CLINICAL TRIAL: NCT00161421
Title: Oral Androgens in Man-3: Pharmacokinetics of Oral Testosterone With Concomitant Inhibition of 5α-Reductase by Dutasteride Short Title: ORAL T-3
Brief Title: Oral Androgens in Man-3 (ORAL T-3) Pharmacokinetics of Oral Testosterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04-4115-D; HD42454; K23HD045386 (NIH); GSK002590
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Contraception; Hypogonadism
Keywords: Male Contraception; Testosterone; Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Leuprolide; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lupron injection at Day -14 with load of dutasteride (24.5 mg) followed by 13 days of Dutasteride. On day 0, 11, 0.5 mg Dutasteride taken daily for next 11 days. Day 1 Oral Testosterone (T) 200mg without food, Day 2 Oral T 400 mg without food, Day 3 Oral T 400 mg with food. During the 2nd week of the study, we will repeat the testosterone doses, with a 2nd formulation of testosterone (Day8, 9, & 10.
  Interventions: Drug: Oral Testosterone; Drug: Leuprolide (Lupron); Drug: Dutasteride

INTERVENTIONS:
Drug: Oral Testosterone — 200 mg (Formulation A) Day 1 400 mg (Formulation A) Day 2, fasting; Day 3, with food 200 mg (Formulation B) Day 8, fasting 400 mg (Formulation B) Day 9, fasting; Day 10, with food
Drug: Leuprolide (Lupron) — 7.5 mg injection into muscle (once) (Day -14)
Drug: Dutasteride — 24.5 mg load (3.5 mg x 7 capsulesDay -14 only) 0.5 mg daily (Day -13 to day -1)
  Other Names: Avodart

SUMMARY:
The purpose of this study is to test the how the body absorbs and processes new forms of oral testosterone. Information gained during the study may help develop better forms of testosterone therapy in the future.

We will be administering three drugs. Dutasteride is FDA approved to treat prostate enlargement. Lupron is approved for treatment of prostate cancer. Testosterone is approved for treatment of testicular insufficiency. They are being used in this study for "off-label" research purposes. This study will allow us to find out the effect of food on two formulations of testosterone taken by mouth, and the relative effect of food on testosterone absorption.

Information from this study may be useful in treatment of men with low testosterone levels and the development of a male hormonal contraceptive.

DETAILED DESCRIPTION:
The drug Lupron, will temporarily turn off the body's production of testosterone after two weeks. At that point, we will administer testosterone by mouth on six days in the next two weeks to see how much is absorbed and present in the bloodstream after administration. The day Lupron is given, and for 24 days after that, subjects will take the second medication, Dutasteride, which alters testosterone breakdown in the body. Fifteen days after the Lupron shot, subjects will take the first formulation of testosterone by mouth and undergo blood draws to see how much of this testosterone makes it into the blood stream and how long it lasts. The next day(Day 2) subjects will take a larger dose of testosterone and undergo blood draws. On study day 3, subjects will again take the larger dose of testosterone, this time with a meal and undergo blood draws. During the 2nd week of the study, subjects will repeat the testosterone doses, with a 2nd formulation of testosterone. The first two doses of testosterone each week will be taken on an empty stomach, while the third will be taken with breakfast. Please note that six study days: 1,2,3,8,9 and 10 will require repeated blood draws over a 12 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Male 18-50 yrs old
* In good general health based on normal screening evaluation (consisting of medical history, physical exam, normal serum chemistry, hematology, and baseline hormone levels)

Exclusion Criteria:

* Poor general health, with abnormal blood results at screening
* A known history of alcohol or drug abuse
* Participation in a long-term male contraceptive study within three months of screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Elevations in serum testosterone | 2 months

SECONDARY OUTCOMES:
Monitoring for any adverse changes in liver function or general health. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: William J Bremner, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Page ST, Bremner WJ, Clark RV, Bush MA, Zhi H, Caricofe RB, Smith PM, Amory JK. Nanomilled oral testosterone plus dutasteride effectively normalizes serum testosterone in normal men with induced hypogonadism. J Androl. 2008 Mar-Apr;29(2):222-7. doi: 10.2164/jandrol.107.002956. Epub 2007 Dec 12. PMID 18077826